CLINICAL TRIAL: NCT01167322
Title: Clinical Study to Assess the Positive Predictive Value of NPC-07 Induced Tissue Fluorescence in Patients With Malignant Glioma (WHO Grades III/IV)
Brief Title: Study of NPC-07 for Fluorescence-guided Resection of Malignant Gliomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NPC-07-1
Record Dates: First submitted 2010-07-16; First posted 2010-07-22 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Malignant Glioma
Keywords: NPC-07, 5-ALA, photodynamic diagnosis, pharmacokinetics
MeSH Terms: conditions — Glioma | interventions — Administration, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NPC-07 (Experimental): Single administration of NPC-07 at a dose of 20mg/kg body weight
  Interventions: Drug: NPC-07 for oral administration

INTERVENTIONS:
Drug: NPC-07 for oral administration — NPC-07, containing 1.5g of 5-aminolevulinic acid hydrochloride per vial, is dissolved in 50 mL of water and will be administered orally 3 hours (range 2-4 hours) prior to induction of anesthesia at a dose of 20mg/kg body weight.
  Other Names: 5-ALA, 5-aminolevulic acid hydrochloride

SUMMARY:
The aim of the present Phase III study is to assess the positive predictive value of NPC-07 (5-aminolevulinic acid hydrochloride) induced tissue fluorescence, safety and pharmacokinetics following a single dose of NPC-07 orally, at a dose of 20mg/kg/body weight, 3 hours prior to induction of anaesthesia for surgery of patients with newly or recurrent malignant glioma (WHO grades III/IV).

Positive predictive value will be confirmed by percentage of patients showing positive tumor cell identification in all biopsies taken from areas of strong and weak fluorescence. This study will be divided into two stages. After reviewing of the result of safety and pharmacokinetics of NPC-07 in small number of subjects by independent safety monitoring committee, more subjects will receive NPC-07 in Step II.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years.
* Radiological suspicion of newly- or recurrent malignant glioma (WHO grades III/IV).
* Indication for surgical tumor resection.
* Karnofsky Performance Score of 60 or higher.
* Provides signed informed consent prior to any study procedures.
* Comply with visit schedule and other rules for patients in study protocol.

Exclusion Criteria:

* Porphyria, hypersensitivity to porphyrins.
* Renal insufficiency: Creatinine 2.0 mg/dL or higher
* Hepatic insufficiency: ALT 100 IU/L or higher, AST 100 IU/L or higher, γ-GTP 100 IU/L or higher or total bilirubin 3 mg/dL or higher
* Chemotherapy or other treatment for other malignant tumors
* Females who are pregnant or potentially childbearing or are breastfeeding
* Participation in other clinical trial in the previous 1 month
* Ineligible patient based on the judgement of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of tissue fluorescence | 1 day
  Positive predictive value of tissue fluorescence defined as the percentage of patients showing positive tumor cell identification in all 6 biopsies taken from areas of strong and weak fluorescence.

SECONDARY OUTCOMES:
Quality of fluorescent tissue | 1 day
  Quality of fluorescent tissue by the judgement of the investigator
Positive predictive value of tissue fluorescence in each biopsy tissue sample | 1 day
  Positive predictive value of tissue fluorescence at the biopsy level defined as the number of tumor positive biopsies among all biopsies taken from areas of strong and weak fluorescence.
Percentage of patients without residual tumor | 3 days
  Percentage of patients without residual tumor in the MRI within 72 hours after surgery
Positive predictive value of non-fluorescent tissue at the biopsy level | 1 day
  Positive predictive value of tissue fluorescence at the biopsy level defined as the number of tumor positive biopsies among the non-fluorescent tissue adjacent to fluorescent tissue areas and the tumor distant cortex with respect to tumor (if available).
Sensitivity as percentage of actual positives and specificity as percentage of actual negatives of fluorescence detection at the biopsy level (if available). | 1 day
  Sensitivity as percentage of actual positives(True positive fraction/True positive fraction + False negative fraction)and specificity as percentage of actual negatives of fluorescence detection (True negative fraction/False positive fraction + True negative fraction) at the biopsy level (if available).
Safety | 28 days
  AEs during study period (Day 0 to Day 28), laboratory parameter, vital signs, EKG, pO2
Pharmacokinetic parameters of NPC-07 and active metabolite (Cmax, AUCt, tmax, t1/2） | 2 days
  Pharmacokinetic parameters of 5-ALA and PPVX (Cmax, AUCt, tmax, t1/2）

CONTACTS AND LOCATIONS:
Overall Officials: Soichiro Shibui, MD, PhD, Study Director — Neurosurgery & Neuro-Oncology Division, National Cancer Center Hospital
Locations (3):
- Japan (3):
  - International Medical Center, Saitama Medical University, Hidaka, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo